CLINICAL TRIAL: NCT05194189
Title: Clinical Efficacy of Megadose Vitamin C in Sepsis (CEMVIS): A Multicenter, Randomized, Single-blind, Placebo-controlled Clinical Trial
Brief Title: Clinical Efficacy of Megadose Vitamin C in Sepsis
Acronym: CEMVIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhanguo, Vice director of the department of critical care medicine, Principal Investigator, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-KY-069-05
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Sepsis; Septic Shock
Keywords: megadose vitamin C
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid; Glucose

STUDY DESIGN:
Intervention Model Description: The participants in treatment group receive intravenous megadose vitamin C. The participants in control group receive 5% glucose injection with same volume.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Megadose vitamin C group (Experimental): 12 g vitamin C (48 ml) will intravenously injected by a infusion pump every 12 h for 4 days or until ICU discharge
  Interventions: Drug: Vitamin C
- Placebo group (Placebo Comparator): 5% glucose solution 48 ml every 12 h for 4 days or until ICU discharge.
  Interventions: Drug: 5% glucose injection

INTERVENTIONS:
Drug: Vitamin C — 12 g vitamin C (48 ml) will be intravenously injected by a infusion pump every 12 h for 4 days or at ICU discharge
  Arms: Megadose vitamin C group
Drug: 5% glucose injection — 5% glucose solution 48 ml every 12 h for 4 days or at ICU discharge.
  Arms: Placebo group

SUMMARY:
In this multicenter, randomized, single-blind, placebo-controlled clinical trial. Patients will be randomly assigned to receive Vitamin C or placebo for 4 days or until ICU discharge (whatever come first). The primary outcome is 28-day all-cause mortality.

DETAILED DESCRIPTION:
Investigational drug: Vitamin C for injection

Study title: Clinical efficacy of megadose vitamin C in sepsis (CEMVIS): A Multicenter, Randomized, Single-blind, Placebo-controlled Clinical Trial

Principal Investigator: Zhanguo Liu, professor, Department of Critical Care Medicine, Zhujiang Hospital, Southern Medical University

Study subjects: Adult septic/septic shock patients with procalcitonin(PCT)≥2ng/ml at recruitment.

Study phase: Investigator Initiated Trial(IIT)

Study objectives: The objective of the study is to determine whether megadose vitamin c, compared to placebo, improve the prognosis of sepsis, including the reduction in mortality, the protection of organ function and reduction of inflammatory response, and to determine the safety of megadose vitamin c in patients with sepsis.

Study design: A Multicenter, Randomized, Single-blind, Placebo-controlled Clinical Trial

Method： Megadose vitamin C group: routine treatment follow the recommendation of the guidelines for sepsis in 2021+ 12 g vitamin C (48 ml) injection every 12 h for 4 days or until ICU discharge (death or transfer from ICU to general ward or discharge), whatever come first. Placebo control group: routine treatment follow the recommendation of the guidelines for sepsis in 2021 + 48ml 5% glucose injection every 12 h for 4 days or until ICU discharge (death or transfer from ICU to general ward or discharge), whatever come first.

Course: 4 days

Sample size: 234

The number of study center: 4

Study center:

1. Department of Critical Care Medicine of Zhujiang Hospital,Guangzhou, Guangdong, China
2. Department of Critical Care Medicine of The First People's Hospital of Foshan, Foshan, Guangdong, China
3. Department of Critical Care Medicine of Dongguan People's Hospital, Dongguan, Guangdong,China
4. Department of Critical Care Medicine of Yunfu People' s Hospital, Yunfu, Guangdong, China
5. Department of Critical Care Medicine of Zhongshan People's Hospital, Zhongshan, Guangdong, China

Primary endpoint: 28-day all-cause mortality.

Secondary endpoints:

1. The state of liver function: the serum level of transaminase(AST、ALT)、total bilirubin at 96 h after randomization
2. The state of lung function: oxygenation index(PaO2/FiO2) at 96h after randomization
3. The state of kidney function: serum level of Creatinine (Cr)、blood urea nitrogen(BUN)、Cystatin(Cys) at 96 h after randomization
4. The state of inflammatory response: the serum level of interleukin-6(IL-6) and C-reactive protein(CRP) at 96 h after randomization.
5. The state of infection: the serum level of procalcitonin(PCT) and white blood cell （WBC） at 96 h after randomization.
6. The state of circulation system: the serum level of lactate at 96 h after randomization
7. Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score at 96 h after randomization
8. The duration of successful cessation of supportive therapies for organ dysfunction including vasoactive agents, mechanical ventilation.
9. The duration of continuous renal replacement therapy(CRRT)
10. The length of stay in ICU

Safety endpoints：

1. adverse events
2. Serious adverse events

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for sepsis-3 developed by the American Society of Critical Care Medicine (SCCM)/European Critical Care Medicine Association (ESICM)
* Age ≥18 years old and age ≤80 years old.
* Procalcitonin ≥2 ng/ml

Exclusion Criteria:

* Age<18 years, or age>80 years.
* Pregnancy or lactating
* A solid-organ or bone marrow transplant patients.
* Patients with myocardial infarction within the past 3 months.
* Advanced pulmonary fibrosis .
* Patients with cardiopulmonary resuscitation before enrollment.
* HIV-positive patients.
* granulocyte-deficient patients.
* blood/lymphatic system tumors are not remission.
* patients with limited care (lack of commitment to full aggressive life support).
* patients with long-term use of immunosuppressive drugs or with immunodeficiency.
* patients with advanced tumors.
* patients combined with non-infectious factors leading to the death(uncontrollable major bleeding, brain hernia, etc.).
* surgically unresolved infection sources(such as some intraperitoneal infection etc.)
* patients allergic to vitamin c.
* patients with G6PD deficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | The outcome will be assessed at the 28 day after enrollment
  All-cause mortality from the enrollment to the 28th days

SECONDARY OUTCOMES:
liver function(1) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the serum level of Alanine transaminase(ALT)
liver function(2) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the serum level of Aspartate transaminase (AST)
liver function(3) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the serum level of total bilirubin
lung function | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  oxygenation index(PaO2/FiO2),the patients treated with extracorporeal membrane oxygenation will not collect this indicator.
kidney function(1) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  serum level of Creatinine (Cr)
kidney function(2) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  serum level of blood urea nitrogen(BUN)
kidney function(3) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  serum level of Cystatin(Cys)
inflammatory response(1) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the serum level of interleukin-6(IL-6)
inflammatory response(2) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the serum level of C-reactive protein(CRP)
Indicators of infection(1) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the serum level of procalcitonin(PCT)
Indicators of infection(2) | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the level of white blood cell count(WBC)
The level of lactate | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  the serum level of lactic acid
Sequential Organ Failure Assessment (SOFA) score | The outcome will be assessed at the 0, 1 ,2 ,4 day after enrollment
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score. SOFA score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. The highest score for each of the six items is 4 points, and the lowest score is 0 points. Finally, the scores of the six items are summed to get the value of the sofa score. The range of the sofa score is 0-24.Higher values represent a worse outcome.
The cessation of mechanical ventilation(MV) administration | The outcome will be assessed at the 28 day after enrollment
  The duration from the MV administration to the successful cessation in hours( The successful cessation is defined as the termination of MV for more than 48-hours. This outcome measure is intended only for patients receiving MV)
The cessation of vasoactive drugs administration | The outcome will be assessed at the 28 day after enrollment
  The duration from the vasoactive drugs administration to the successful cessation in hours( The successful cessation is defined as the attainment of a clinician-prescribed mean arterial pressure target for more than 24-hours without the use of vasoactive drugs.This outcome measure is intended only for patients receiving vasoactive drugs)
The duration of CRRT | The outcome will be assessed at the 28 day after enrollment
  The duration of CRRT therapy in hours( This outcome measure is intended only for patients receiving CRRT)
ICU length of stay | The outcome will be assessed at the 28 day after enrollment
  ICU length of stay

OTHER OUTCOMES:
Incidence of adverse events | The outcome will be assessed at the 28 day after enrollment
  A adverse event refers to any adverse medical event that occur after the intervention of trial. The adverse events are not necessarily causally related to the trial treatment.
Incidence of serious adverse events | The outcome will be assessed at the 28 day after enrollment
  Any adverse medical event occurs at any dose that meets one or more of the following criteria: 1. causes death 2.life-threatening 3. requires hospitalization or hospitalization for an extended period of time 4. causes permanent or significant disability and functional defects 5. causes deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Liu, M.D.PhD, Principal Investigator — Department of Critical Care Medicine of Zhujiang Hospital
Locations (4):
- China (4):
  - Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University, Guanzhou, Guangdong
  - Department of Critical Care Medicine of Yunfu People's Hospital, Yunfu, Guangdong
  - Department of Critical Care Medicine of Zhongshan People's Hospital, Zhongshan, Guangzhou
  - Department of Critical Care Medicine of Nanfang Hospital of Southern Medical University, Guanzhou

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analyzed during the study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Liu F, Zhu Y, Zhang J, Li Y, Peng Z. Intravenous high-dose vitamin C for the treatment of severe COVID-19: study protocol for a multicentre randomised controlled trial. BMJ Open. 2020 Jul 8;10(7):e039519. doi: 10.1136/bmjopen-2020-039519. PMID 32641343
- [Background] Chang P, Liao Y, Guan J, Guo Y, Zhao M, Hu J, Zhou J, Wang H, Cen Z, Tang Y, Liu Z. Combined Treatment With Hydrocortisone, Vitamin C, and Thiamine for Sepsis and Septic Shock: A Randomized Controlled Trial. Chest. 2020 Jul;158(1):174-182. doi: 10.1016/j.chest.2020.02.065. Epub 2020 Mar 31. PMID 32243943